CLINICAL TRIAL: NCT05754671
Title: PERCEPTUAL EVALUATION OF THE TRACHEO-OESOPHAGEAL VOICE: ITALIAN VALIDATION OF THE SUNDERLAND TRACHEOESOPHAGEAL PERCEPTUAL SCALE (I-SToPS)
Brief Title: Perceptual Assessment of the Tracheoesophageal Voice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D'Alatri Lucia, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3554
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Tracheo-Esophageal Fistula Following Tracheostomy
Keywords: voice prosthesis; perceptual evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laryngectomized patients (Experimental)
  Interventions: Other: voice recording
- health professionals (Experimental)
  Interventions: Other: perceptual assessment of the recorded voice sample

INTERVENTIONS:
Other: perceptual assessment of the recorded voice sample — perceptual assessment of the recorded voice samples
  Arms: health professionals
Other: voice recording — voice recording
  Arms: laryngectomized patients

SUMMARY:
Aim of this study was to validate the Sunderland Tracheoesophageal Perceptual Scale (SToPS) in Italian language by checking the inter- and intra-rater reliability.

The validation of the tool involved the following steps: 1) Translation and adaptation of the SToPS into Italian language; 2) Recruitment of participants (43 laryngectomized patients with a voice prosthesis and 12 health professionals - 6 speech and language therapists (SLTs) and 6 Ear, Nose, and Throat (ENTs) surgeons - classified into experienced or not at assessing voice; 3) Recording of patients' speech samples; 4) Perceptual evaluation of recorded speech samples (test and re-test) performed by the 12 health professionals; 5) Statistical analysis (quadratic weighted Cohen Kappa and weighted Kappa of Light coefficients).

SLTs with specific experience in tracheo-esophageal and laryngeal voice rated more reliably than the others raters. For all groups of raters, the inter-rater agreement was worse than the intra-rater one for 9/10 parameters. Exclusively for experienced SLTs, only the "Impairment of social acceptability" parameter reached a good level of inter-rater agreement.

In conclusion, the Italian version of SToPS can be considered a reliable tool. As in the original version, expert SLTs may be considered the optimal judges for tracheoesophageal voice assessment.

ELIGIBILITY:
Inclusion Criteria:

* native Italian speakers;
* ability to produce TE voice.

Exclusion Criteria:

* reading difficulties;
* presence or suspicion of disease recurrence;
* other communication problems not related to Total laryngectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Reliability | 4 months
  The primary aim of this study was to carry out a psychometric validation in Italian of a perceptual evaluation scale for use by clinicians. The intra- and inter-rater reliability of each parameter was analyzed with Cohen's kappa weighted quadratic statistic.
  A weighted average kappa coefficient equal to or greater than 0.61 has been considered a "good" level of agreement.

SECONDARY OUTCOMES:
Training | 4 months
  Secondary aim was to investigate whether the SToPS could be used without training, using written guidelines only and focusing on the effect of experience on the administration of the SToPS. For this reason, the reliability results obtained were compared with those of the original study.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia D'Alatri, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No